CLINICAL TRIAL: NCT04012125
Title: The Effect of Flexible Thoracolumbar Brace on Scoliosis in Cerebral Palsy, Prospective, Randomized, Open-label Trial
Brief Title: The Effect of Flexible Thoracolumbar Brace on Scoliosis in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B-1805/471-003
Record Dates: First submitted 2019-06-05; First posted 2019-07-09 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Brace; Scoliosis
MeSH Terms: conditions — Cerebral Palsy; Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective, single-arm trial (Experimental)
  Interventions: Device: flexible thoracolumbar brace

INTERVENTIONS:
Device: flexible thoracolumbar brace — Subjects would wear the flexible thoracolumbar brace over 18 hours a day

SUMMARY:
The Effect of Flexible Thoracolumbar Brace on Scoliosis in Cerebral Palsy, Prospective, Randomized, Open-label Trial

ELIGIBILITY:
Inclusion Criteria:

* GMFCS level III, IV, V of the Cerebral palsy
* 20-45 degree of Cobb's angle

Exclusion Criteria:

* less than 20 degree or more than 45 degree of Cobb's angle
* Neuromuscular disease including congenital myopathy, spinal muscular atrophy, muscular dystrophy and poliomyelitis
* Acute lumbar pain
* Fixed scoliosis

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Change of scoliosis | 6months
  Cobb's angle in the whole spine anteroposterior view of X-ray, before and immediately after, and 6months after wearing FLEXpine brace

SECONDARY OUTCOMES:
Pain of the back (thorax) | 6 months
  Patients check the scale through the visual analog scale
change of quality of life (aspect of the parents) | 6 months
  Parent of the patients assessed "caregiver experience with neuromuscular disease" before and 6-month after wearing FLEXpine brace

CONTACTS AND LOCATIONS:
Overall Officials: JUSEOK RYU, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul national university bundang hospital, Seongnam-si, Bundang-gu, South Korea

IPD SHARING:
Plan to Share IPD: No